CLINICAL TRIAL: NCT05895097
Title: Impact of Conduction System Pacing on Left Ventricular Remodeling After Transcatheter Aortic Valve Implantation
Brief Title: Conventional Versus Left Bundle Branch Pacing in TAVI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Klemen Steblovnik, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACE TAVI
Record Dates: First submitted 2023-02-06; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Stenosis; Heart Failure; Pacemaker-Induced Cardiomyopathy; Transcatheter Aortic Valve Implantation
Keywords: Transcatheter Aortic Valve Implantation; Left bundle branch pacing
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional pacing (Active Comparator)
  Interventions: Device: Conventional pacing
- LBB pacing (Experimental)
  Interventions: Device: Left bundle branch pacemaker

INTERVENTIONS:
Device: Left bundle branch pacemaker — Left bundle branch pacing (LBBP) will be the pacing technique. In brief, after localizing the His bundle area the LBBP lead will be positioned approximately 1-1.5 cm distal to the His bundle position in the right ventricular septum. Before screwing the lead deep into the interventricular septum, the suitable position will be confirmed by fluoroscopic signs and adequate paced QSR morphology. Final lead position will be confirmed according to ECG parameters. Given that the pacing parameters with LBBP are typically low and stable, backup RV lead will not be mandatory.
  Arms: LBB pacing
Device: Conventional pacing — Right ventricular pacing in patients with LVEF ≥ 40% and cardiac resynchronization therapy in patients with LVEF < 40 %
  Arms: Conventional pacing

SUMMARY:
This randomized study compares the effects of conventional (right ventricular pacing in patients with LVEF ≥ 40% and cardiac resynchronization therapy in patients with LVEF < 40 %) versus left bundle branch pacing on left ventricular remodelling in patients with reduced left ventricular ejection fraction (< 50 %) that need permanent pacemaker implantation after transcatheter aortic valve implantation (TAVI).

DETAILED DESCRIPTION:
Bradycardic heart rhythm disturbances are a common complication of TAVI. Patients who will develop the indication for permanent pacemaker implantation after TAVI will be randomly assigned to either the experimental (left bundle branch pacing) or conventional (right ventricular pacing in patients with LVEF ≥ 40% and cardiac resynchronization therapy in patients with LVEF < 40 %) group. The investigators will compare the left ventricular ejection fraction (primary outcome) 12 months after randomization. The investigators will also compare electrocardiographic (QRS duration), clinical (NYHA status, 6-minute walking test, handgrip test, Kansas City Cardiomyopathy Questionnaire) and laboratory (proBNP) parameters 6 and 12 months, and other echocardiographic (left ventricular systolic and diastolic diameter, signs of dyssynchrony, myocardial work) parameters 12 months after pacemaker implantation in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Indication for permanent pacemaker implantation after transcatheter aortic valve implantation (during the same hospitalization)
* Left ventricular ejection fraction < 50 %.

Exclusion Criteria:

* Unsuccessful TAVI procedure with life expectancy < 1 year
* Ischemic cardiomyopathy with interventricular septal fibrosis (at least echocardiographic signs of fibrosis)
* Severe kidney failure (glomerular filtration rate < 30 ml/min)
* Previous permanent pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 12 months

SECONDARY OUTCOMES:
Left ventricular systolic diameter | 12 months
Left ventricular diastolic diameter | 12 months
Global work index | 12 months
  Amount of myocardial work performed by the left ventricle during systole.
Global constructive work | 12 months
  Positive work performed in systole + negative work performed in isovolumetric relaxation
Global wasted work | 12 months
  Negative work performed in systole + positive work performed in isovolumetric relaxation
Global work efficiency | 12 months
  Percentage of constructive work over total work = Constructive work/(constructive work + wasted work)
Signs of mechanical dyssynchrony | 12 months
  Presence of at least one of the echocardiographic signs of mechanical dyssynchrony, such as apical rocking and septal flash.
Systolic pulmonary artery pressure (echocardiographic parameter) | 12 months
NT-proBNP concentration | 6 and 12 months
NYHA status | 6 and 12 months
6-minute walking test | 6 and 12 months
Hand grip test | 6 and 12 months
The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 6 and 12 months
  KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
QRS duration | baseline, 6, and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided